CLINICAL TRIAL: NCT01103349
Title: Randomised, Double Blind, Double Dummy, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of 6 Weeks of Oral BI 671800 ED Twice Daily (b.i.d.), Montelukast Once Daily (q.d.) or Placebo in Symptomatic Asthmatic Patients on Low Dose Fluticasone Propionate MDI (Metered Dose Inhaler)
Brief Title: BI 671800 in Asthmatic Patients on Inhaled Corticosteroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1268.16; 2009-014551-80 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-03-19; First posted 2010-04-14 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — BI 671800; montelukast

ARMS (3):
- BI 671800 (Experimental): Patients receive BI 671800 capsules twice daily
  Interventions: Drug: BI 671800
- Montelukast (Active Comparator): Patients receive Montelukast encapsulated tablets once daily
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Patients receive placebo capsules and/or encapsulated placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 671800 — Double blind randomised parallel group study to assess efficacy and tolerability of BI 617800 in patients with symptomatic asthma
  Arms: BI 671800
Drug: Placebo — Patients receive placebo capsules and/or encapsulated tablets
  Arms: Placebo
Drug: Montelukast — Double blind randomised parallel group study to assess efficacy and tolerability of BI 671800 in patients with symptomatic asthma
  Arms: Montelukast

SUMMARY:
This is a 6 week study to assess the effect of BI 671800 in patients with asthma. It is a double blind, parallel arm trial testing the safety and efficacy of BI 671800. The main objective is to assess the effect on lung function. The study will also provide data on the pharmacokinetics of BI 671800.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent consistent with ICH-GCP
2. Three month history of reversible (12% and 200 mL in forced expiratory volume in one second - FEV1) asthma (according to GINA) with following spirometry at randomisation: FEV1 60%- 85%.
3. Stable inhaled corticosteroids (iCS) dose 3 months prior to screening.
4. Diagnosis of asthma prior to 40 years.
5. Asthma Control Questionnaire (ACQ) at least 1.5 at randomisation.
6. Male or female 18 to 65 years.
7. Non-smokers or ex-smokers (less than 10 pack years history) with negative cotinine screen.
8. Able to perform pulmonary function testing.

Exclusion criteria:

1. Significant diseases other than asthma or allergic rhinitis.
2. Hepatic transaminases or total bilirubin greater than 1.5 ULN.
3. Hospitalisation for asthma exacerbation or asthma related intubation within 3 months.
4. Uncontrolled asthma on iCS + other controller.
5. Respiratory tract infection or exacerbation within 4 weeks.
6. FEV1 less than 40%, more than 12 puffs rescue salbutamol on more than two consecutive days, or asthma exacerbation during run-in period.
7. Participation in another interventional study.
8. Pregnant or nursing women.
9. Women of child bearing potential not using appropriate methods of birth control as defined by the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-04-20 (Actual); Primary Completion 2011-08-09 (Actual); Study Completion 2011-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- United States (6):
  - 1268.16.01004 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1268.16.01001 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1268.16.01006 Boehringer Ingelheim Investigational Site, Plymouth, Minnesota
  - 1268.16.01003 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1268.16.01002 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1268.16.01005 Boehringer Ingelheim Investigational Site, El Paso, Texas
- 1268.16.43002 Boehringer Ingelheim Investigational Site, Feldbach, Austria
- Germany (18):
  - 1268.16.49018 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1268.16.49014 Boehringer Ingelheim Investigational Site, Bamberg
  - 1268.16.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1268.16.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1268.16.49010 Boehringer Ingelheim Investigational Site, Berlin
  - 1268.16.49012 Boehringer Ingelheim Investigational Site, Berlin
  - 1268.16.49013 Boehringer Ingelheim Investigational Site, Berlin
  - 1268.16.49016 Boehringer Ingelheim Investigational Site, Berlin
  - 1268.16.49008 Boehringer Ingelheim Investigational Site, Erfurt
  - 1268.16.49005 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1268.16.49015 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1268.16.49011 Boehringer Ingelheim Investigational Site, Hamburg
  - 1268.16.49009 Boehringer Ingelheim Investigational Site, Hanover
  - 1268.16.49017 Boehringer Ingelheim Investigational Site, Hanover
  - 1268.16.49007 Boehringer Ingelheim Investigational Site, Koblenz
  - 1268.16.49006 Boehringer Ingelheim Investigational Site, Lübeck
  - 1268.16.49002 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1268.16.49003 Boehringer Ingelheim Investigational Site, Weinheim
- Italy (4):
  - 1268.16.39006 Boehringer Ingelheim Investigational Site, Ferrara
  - 1268.16.39007 Boehringer Ingelheim Investigational Site, Milan
  - 1268.16.39004 Boehringer Ingelheim Investigational Site, Pietra Ligure (SV)
  - 1268.16.39001 Boehringer Ingelheim Investigational Site, Pisa
- New Zealand (2):
  - 1268.16.64001 Boehringer Ingelheim Investigational Site, Christchurch NZ
  - 1268.16.64003 Boehringer Ingelheim Investigational Site, Greenlane East Auckland
- South Korea (10):
  - 1268.16.82008 Boehringer Ingelheim Investigational Site, Anyang
  - 1268.16.82009 Boehringer Ingelheim Investigational Site, Bucheon-si
  - 1268.16.82007 Boehringer Ingelheim Investigational Site, Cheongju-si
  - 1268.16.82006 Boehringer Ingelheim Investigational Site, Daegu
  - 1268.16.82010 Boehringer Ingelheim Investigational Site, Gwangju
  - 1268.16.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.16.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.16.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.16.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1268.16.82003 Boehringer Ingelheim Investigational Site, Suwon
- Sweden (3):
  - 1268.16.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1268.16.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1268.16.46003 Boehringer Ingelheim Investigational Site, Örebro
- Turkey (Türkiye) (5):
  - 1268.16.90002 Boehringer Ingelheim Investigational Site, Bursa
  - 1268.16.90003 Boehringer Ingelheim Investigational Site, Istanbul
  - 1268.16.90004 Boehringer Ingelheim Investigational Site, Istanbul
  - 1268.16.90006 Boehringer Ingelheim Investigational Site, Istanbul
  - 1268.16.90001 Boehringer Ingelheim Investigational Site, Mersin
- United Kingdom (4):
  - 1268.16.44005 Boehringer Ingelheim Investigational Site, Chertsey
  - 1268.16.44004 Boehringer Ingelheim Investigational Site, London
  - 1268.16.44002 Boehringer Ingelheim Investigational Site, Manchester
  - 1268.16.44003 Boehringer Ingelheim Investigational Site, Southampton

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIa, multicentre, multinational, randomised, double-blind, double-dummy, placebo-controlled, parallel group study to assess the efficacy and safety of oral BI 671800 ED 400 mg b.i.d., montelukast 10 mg q.d., or placebo in symptomatic asthma patients on Fluticasone propionate Hydrofluoralkane Metered Dose Inhaler (100μg b.i.d.).
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all subjects as required.
Groups:
- Placebo: Daily treatment with 4 oral capsules of BI 671800 Ethylenediamine (ED) placebo in the morning and 4 oral capsules of BI 671800 ED placebo plus 1 over-encapsulated montelukast placebo tablet in the evening, for a total treatment period of 6 weeks.
- BI 671800 400 mg Bid: Daily treatment with 4 oral capsules of 100 milligram (mg) BI 67800 Ethylenediamine (ED) in the morning and 4 oral capsules of 100 mg BI 67800 ED plus 1 over-encapsulated montelukast placebo tablet in the evening, for a total treatment period of 6 weeks.
- Montelukast 10 mg qd: Daily treatment with 4 oral capsules of BI 67800 Ethylenediamine (ED) Placebo in the morning and 4 oral capsules of BI 67800 ED Placebo plus 1 table of 10 mg over-encapsulated montelukast in the evening, for a total treatment period of 6 weeks.
Period: Overall Study
Arm/Group | Placebo | BI 671800 400 mg Bid | Montelukast 10 mg qd
Started | 95 | 81 | 67
Completed | 84 | 74 | 63
Not Completed | 11 | 7 | 4
Not completed — Adverse Event | 8 | 5 | 3
Not completed — Consent withdrawn | 1 | 0 | 0
Not completed — Incorrectly included in the trial | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — did not want to take trial medication | 0 | 1 | 0
Not completed — forgot to take medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All randomized patients who received at least one dose of treatment, the treated set was used in the safety analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 671800 400 mg Bid | Montelukast 10 mg qd | Total
Number analyzed (Participants) | 95 | 81 | 67 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.64) | 41.8 (12.67) | 41.7 (11.97) | 41.6 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 50 | 42 | 147
  Male | 40 | 31 | 25 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 2 | 8
  Not Hispanic or Latino | 93 | 77 | 65 | 235
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 12 | 6 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 77 | 66 | 56 | 199
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 3 | 11
Percentage of predicted forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: Percentage of predicted FEV1] | 68.089 (10.9109) | 69.286 (10.5542) | 69.842 (10.5288) | 68.986 (10.6644)

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) % Predicted Trough Change From Baseline (Mean Observed in the 2 Weeks Prior to Treatment) After Six Weeks of Treatment
Description: Forced expiratory volume in one second (FEV1) % predicted trough change from baseline (mean observed in the 2 weeks prior to treatment) after 6 weeks of treatment, where trough FEV1 % predicted was defined as the mean of the FEV1 % predicted trough values at 25 minutes and 10 minutes prior to dosing on clinic visit.
  MMRM in the statistical test comments is Mixed effects model with repeated measures.
Time Frame: Measurements at baseline (mean observed in the 2 weeks prior to treatment) and at week 6 of treatment.
Population: Statistical analysis was performed on randomized patients who received at least one dose of treatment and had both baseline and the post-baseline measurement at 6 weeks for the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: FEV1 percent predicted
Arm/Group | Placebo | BI 671800 400 mg Bid | Montelukast 10 mg qd
Number analyzed (Participants) | 81 | 74 | 62
FEV1 percent predicted | -0.859 (1.029) | 3.011 (1.082) | 1.510 (1.181)
Statistical Analysis 1: Comparison: Placebo vs BI 671800 400 mg Bid; H0: Mean FEV1 % predicted trough change from baseline (BI671800 ED 400 mg bid) ≤ Mean FEV1 % predicted trough change from baseline (placebo); Test type: Superiority; p = 0.0050, Mixed Models Analysis — α=0.025 one-sided; MMRM with baseline, treatment, day, treatment by day interaction and baseline by day interaction as fixed effects and patient as a random effect; Adjusted mean treatment differences = 3.870, 95% CI 2-sided [0.931 to 6.809], Standard Deviation 1.494
Statistical Analysis 2: Comparison: Placebo vs Montelukast 10 mg qd; H0: Mean FEV1 % predicted trough change from baseline (Montelukast 10 mg qd) ≤ Mean FEV1 % predicted trough change from baseline (placebo); Test type: Superiority; p = 0.0657, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 2.369, 95% CI [-0.713 to 5.452], Standard Deviation 1.567
Statistical Analysis 3: Comparison: BI 671800 400 mg Bid vs Montelukast 10 mg qd; H0: Mean FEV1 % predicted trough change from baseline (BI671800 ED 400 mg bid) ≤ Mean FEV1 % predicted trough change from baseline (Montelukast 10 mg qd); Test type: Superiority; p = 0.1748, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = 1.501, 95% CI 2-sided [-1.652 to 4.653], Standard Deviation 1.602

2. Secondary Outcome: Asthma Control Questionnaire (ACQ) Mean Change in Score on a Scale From Baseline After Six Weeks of Treatment
Description: Asthma Control Questionnaire (ACQ) mean score change from baseline (mean ACQ score obtained at Week 0) after six weeks of treatment.
  The Asthma Control Questionnaire (ACQ) is a patient-reported outcome questionnaire containing 7 items. The items are equally weighted and the ACQ score is the mean of the 7 items and therefore between 0 (well controlled) and 6 (extremely poorly controlled) These questions based on recall of the previous 7 days comprise breathlessness, nocturnal waking, symptoms on waking, activity limitation, wheeze, frequency of Short-acting beta-adrenergic (SABA) use, and categorized pre-bronchodilator FEV1% predicted.
Time Frame: Measurements at baseline (mean ACQ score obtained at Week 0) and at week 6 of treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | BI 671800 400 mg Bid | Montelukast 10 mg qd
Number analyzed (Participants) | 81 | 74 | 62
Score on a scale | -0.418 (0.081) | -0.698 (0.085) | -0.598 (0.093)
Statistical Analysis 1: Comparison: Placebo vs BI 671800 400 mg Bid; Test type: Superiority; p = 0.0092, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -0.280, 95% CI 2-sided [-0.512 to -0.048], Standard Deviation 0.118
Statistical Analysis 2: Comparison: Placebo vs Montelukast 10 mg qd; Test type: Superiority; p = 0.0732, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -0.180, 95% CI 2-sided [-0.423 to 0.063], Standard Deviation 0.124
Statistical Analysis 3: Comparison: BI 671800 400 mg Bid vs Montelukast 10 mg qd; Test type: Superiority; p = 0.2139, Mixed Models Analysis — α=0.025 one-sided; [statistical method as in outcome 1, analysis 1]; Adjusted mean treatment differences = -0.100, 95% CI 2-sided [-0.347 to 0.147], Standard Deviation 0.126

ADVERSE EVENTS:
Time Frame: Adverse Events: Day of the first dose till the day of the last dose + 5 days residual effect period, up to 64 days. All-Cause Mortality: Day of the first dose till the day of the last dose + 2 weeks follow up, up to 73 days.
Description: Treated Set (TS): All randomized patients who received at least one dose of treatment, the treated set was used in the safety analysis.
Arm/Group | Placebo | BI 671800 400 mg Bid | Montelukast 10 mg qd
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/81 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/95 | 1/81 | 0/67
Other Adverse Events (participants affected / at risk) | 18/95 | 10/81 | 8/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | BI 671800 400 mg Bid (N=81) | Montelukast 10 mg qd (N=67)
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | BI 671800 400 mg Bid (N=81) | Montelukast 10 mg qd (N=67)
Nasopharyngitis (Infections and infestations) | 5 | 5 | 3
Headache (Nervous system disorders) | 5 | 4 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.